CLINICAL TRIAL: NCT05608200
Title: Lenvatinib, Sintilimab Plus TACE Versus Lenvatinib Plus TACE for Patients With Advanced Hepatocellular Carcinoma: a Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Lenvatinib+Sintilimab+TACE vs. Lenvatinib+TACE for Advanced HCC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-10
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Hepatocellular Carcinoma; Lenvatinib; Sintilimab; Transarterial Chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Len-Sin-TACE (Experimental): Lenvatinib, Sintilimab Plus TACE
  Interventions: Drug: Lenvatinib, sintilimab plus TACE
- Len-TACE (Active Comparator): Lenvatinib Plus TACE
  Interventions: Drug: Lenvatinib plus TACE

INTERVENTIONS:
Drug: Lenvatinib, sintilimab plus TACE — Lenvatinib 12mg (body weight ≥60kg) or 8mg (body weight <60kg) P.O. qd and sintilimab (200mg I.V. q3w) will be started at 3-7 days after the first TACE. TACE will be repeated if clinically indicated. Treatment of sintilimab will last up to 24 months. Patients will be allowed to have lenvatilib or sintilimab as a sigle agent and will be still considered on study when the other drug cause intolerable toxicity.
  Arms: Len-Sin-TACE
Drug: Lenvatinib plus TACE — Lenvatinib 12mg (body weight ≥60kg) or 8mg (body weight <60kg) P.O. qd will be started at 3-7 days after the first TACE. TACE will be repeated if clinically indicated. The interruption, dose reduction and discontinuation of lenvatinib depended on the presence and severity of toxicities according to the drug directions.
  Arms: Len-TACE

SUMMARY:
This study is conducted to evaluate the efficacy and safety of lenvatinib, sintilimab plus TACE (Len-Sin-TACE) compared with lenvatinib plus TACE (Len-TACE) for patients with advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
This is a multicenter, prospective and randomized controlled trial to evaluate the efficacy and safety of Len-Sin-TACE versus Len-TACE for patient with advanced HCC.

427 patients with advanced HCC (CNLC IIIa-IIIb/BCLC C stage) will be enrolled in this study. The patients will receive either Len-Sin or Len alone after first TACE using an 2:1 randomization scheme. In the Len-Sin arm, lenvatinib 12mg (body weight ≥60kg) or 8mg (body weight <60kg) P.O. qd and sintilimab (200mg I.V. q3w) will be started at 3-7 days after the first TACE. In the the Len arm, lenvatinib 12mg (body weight ≥60kg) or 8mg (body weight <60kg) P.O. qd will be started at 3-7 days after the first TACE.

TACE will be repeated if clinically indicated based on the evaluation of follow-up laboratory and imaging examination. Lenvatinib will last until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. Sintilimab will last up to 24 months, or until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. In the Len-Sin arm, patients will be allowed to have lenvatinib or sintilimab as a sigle agent and will be still considered on study when the other drug cause intolerable toxicity.

The primary end point of this study is overall survival (OS). The secondary endpoints are progression-free survival (PFS), time to progression (TTP), objective response rate (ORR), disease control rate (DCR), and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Advanced HCC (BCLC stage C, or CNLC IIIa and IIIb ) with diagnosis confirmed by histology/cytology or clinically
* Patients who have Tumor recurrence after surgical resection or ablation are allowed to be included
* At least one measurable intrahepatic target lesion
* Child-Pugh class A/B
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 3 months

Exclusion Criteria:

* Obstructive portal vein tumor thrombus involving both the left and right portal vein or main portal vein without collateral vessels
* Vascular invasion involving inferior vena cava
* Central nervous system metastasis
* Patients who received prior systemic therapy, immunotherapy, TACE, transcatheter arterial radioembolization (TARE), transcatheter arterial embolization (TAE), hepatic arterial infusion chemotherapy (HAIC) or radiation therapy for HCC
* History of organ and cell transplantation
* History of bleeding from esophageal and gastric varices
* History of hepatic encephalopathy
* hematologic examination: white blood cell count <3.0×10^9/L, platelets <50×10^9/L
* Prothrombin time prolongation ≥ 4s
* Severe organ (heart, lung, kidney) dysfunction
* History of malignancy other than HCC
* Active hepatitis B or C infection; hepatitis B virus (HBV) DNA > 1000 copies/ml; hepatitis C virus (HCV) RNA > 1000 copies/ml. Those who possess the indicators lower than the above criteria after nucleotide antiviral treatment can be enrolled

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 4 years
  The time from date of randomization to death due to any cause.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 4 years
  The time from date of randomization until the first occurrence of disease progression (according to mRECIST) or death due to any cause, whichever occurs first.
Time to Progression (TTP) | 4 years
  The time from date of randomization until the first occurrence of disease progression (according to mRECIST).
Objective response rate (ORR) | 4 years
  The proportion of patients with the best response of complete response (CR) or partial response (PR) according to mRECIST.
Disease control rate (DCR) | 4 years
  The proportion of patients with the best response of CR, PR, or stable disease (SD) according to mRECIST.
Adverse Events (AEs) | 4 years
  Number of patients with AEs assessed by Common Terminology Criteria for Adverse Events v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Kangshun Zhu, MD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China